CLINICAL TRIAL: NCT03179462
Title: "Ounce-equivalents" in the Protein Foods Group: Benefits of Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 206579
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Results first posted 2021-09-30 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-10

CONDITIONS: Protein Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pork intake (Experimental): Subjects will consume 2 ounces of cooked lean pork following diet normalization for 3 days.
  Interventions: Dietary Supplement: Pork intake
- Mixed nuts intake (Experimental): Subjects will consume 1 ounce of mixed nuts following diet normalization for 3 days.
  Interventions: Dietary Supplement: Mixed nuts intake
- Tofu intake (Experimental): Subjects will consume 2 ounces of tofu following diet normalization for 3 days.
  Interventions: Dietary Supplement: Tofu intake

INTERVENTIONS:
Dietary Supplement: Pork intake — Each participant will consume 2 ounces of cooked lean pork.
  Arms: Pork intake
Dietary Supplement: Mixed nuts intake — Each participant will consume 1 ounce of mixed nuts.
  Arms: Mixed nuts intake
Dietary Supplement: Tofu intake — Each participant will consume 2 ounces of tofu.
  Arms: Tofu intake

SUMMARY:
The investigators will examine the effects of a given amount of a protein food source such as pork, mixed nuts, and tofu on anabolic response at the whole body and muscle levels in young, healthy adults.

DETAILED DESCRIPTION:
Over the past 35 years the United States Department of Agriculture (USDA) Dietary Guidelines for Americans (DGAs) has sought to translate recommendations on nutrient requirements (i.e., Recommended Dietary Allowances) from the Food and Nutrition Board of the Institute of Medicine (IOM) into practical nutritional advice for the American public. Although the DGAs are intended to incorporate additional scientific evidence, the lack of appropriate focus on protein nutrition is a major shortcoming of the DGAs. Not only is the amount of protein not a major focus, absolutely no mention is made of protein quality. In general, animal proteins have much higher the Digestible Indispensable Amino Acid Scores (DIAASs) than plant proteins, often by as much as two fold. Account has not been taken of DIAAS, or even the general concept of the importance of the amount and profile of essential amino acids in individual proteins, in formulation of MyPlate or the scientific report of the DGAs Committee. This is because a classification does not apply to most plant proteins, despite the fact that in the IOM report stating the Recommended Dietary Allowance for protein it is specified that this refers to "high quality protein. To help the consumer meet protein needs while achieving the goal of varied protein food sources, the DGAs Committee published "ounce equivalents" in the protein foods group. It is stated among other equivalents cited, that 1 ounce (oz.) of meat is equivalent to 1 tablespoon (Tbsp.) of peanut butter and 1/4 cup (0.5 ounces) of cooked kidney beans. But are they really equivalent? This indicates that the "ounce equivalents" of protein foods in MyPlate are not equivalent in any parameter that might be used to assess nutritional benefit, and demonstrates that the bias against animal proteins is in the Dietary Guidelines. The misrepresentation of the equivalencies of various food sources of protein in MyPlate raises the question of the process by which this occurred, and how can the process be influenced to more accurately reflect that high quality of animal proteins? Therefore, developing convincing data to correct the MyPlate "ounce equivalents" of protein foods is an achievable goal. In general, dietary protein intake serves many physiological roles, but the most prominent is the maintenance or gain of body protein. This is accomplished by stimulation of protein synthesis, the inhibition of protein breakdown, or a combination. Thus, the functional response to consumption of a given amount of a protein food source is best assessed by quantifying the rates of protein synthesis and breakdown at the whole body level as well as at the muscle level in order to calculate the anabolic response. The investigators propose to make these measurements in response to intake of "equivalent "(according to MyPlate) amounts of pork, mixed nuts and tofu. Moreover, the functional responses to these varied sources of protein we will examine coincide with the predictions from the USDA nutrient data base, and calculation of the DIAAS will provide needed support to redefine "ounce equivalents" of protein food sources according to those data bases for all animal and plant sources of protein.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18-40 years
* BMI from 20 to 29.9 kg/m2

Exclusion Criteria:

* Current diagnosis of diabetes
* History of malignancy in the 6 months prior to enrollment
* History of a chronic inflammatory condition or other chronic diseases (Lupus, HIV/AIDS, etc)
* History of weight reduction surgery (Lapband, gastric sleeve, etc.)
* Pregnant females
* Subjects who do not or will not eat animal proteins
* Subjects allergic to pork, tree or peanuts, or soybeans
* Subjects who cannot refrain from consuming protein or amino acid supplements during their participation in this study
* Subjects who report regular resistance training exercise > one per week
* Hemoglobin < 9.5 g/dL at the screening visit
* Platelets < 250,000 at the screening visit
* Concomitant use of corticosteroids (ingestion, injection or transdermal)
* Any other disease or condition that would place the subject at increased risk of harm if they were to participate, at the discretion of the study physician

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pork Intake | Mixed Nuts Intake | Tofu Intake
Started | 9 | 10 | 8
Completed | 8 | 8 | 8
Not Completed | 1 | 2 | 0
Not completed — screening failure | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pork Intake | Mixed Nuts Intake | Tofu Intake | Total
Number analyzed (Participants) | 9 | 10 | 8 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 8 | 27
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 4 | 14
  Male | 5 | 4 | 4 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 7 | 7 | 7 | 21
  Black/African American | 2 | 2 | 1 | 5
  Asian | 0 | 1 | 0 | 1
  Other Race | 0 | 0 | 0 | 0
  Hispanic ethnicity | 0 | 1 | 0 | 1
  non-Hispanic ethnicity | 9 | 9 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Net Protein Synthesis Rate
Description: Net protein synthesis rate is determined in the 4.5-hours basal fasted period and 4-hours post-meal period over the 8.5-hour experimental period.
Time Frame: Change from 4.5 to 8.5 hours.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Pork Intake | Mixed Nuts Intake | Tofu Intake
Number analyzed (Participants) | 8 | 8 | 8
grams | 8.65 (1.6) | 1.97 (1.04) | 5.69 (0.54)
Statistical Analysis 1: Comparison: Pork Intake vs Mixed Nuts Intake vs Tofu Intake; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a subject enrolled through their last study visit (e.g. 1 month more or less).
Arm/Group | Pork Intake | Mixed Nuts Intake | Tofu Intake
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT03179462/Prot_SAP_000.pdf